CLINICAL TRIAL: NCT03703466
Title: An Open-Label, Randomized Phase 2 Study of the Impact of Food on Tolerability When Receiving Abemaciclib for Patients With Previously Treated Hormone Receptor-Positive, HER2-Negative, Metastatic Breast Cancer
Brief Title: A Study of Abemaciclib (LY2835219) With and Without Food in Participants With Metastatic Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 17041; I3Y-MC-JPCP (Other: Eli Lilly and Company); 2018-001853-28 (EudraCT Number)
Record Dates: First submitted 2018-10-05; First posted 2018-10-12 (Actual); Results first posted 2020-08-13 (Actual); Last update posted 2024-04-02 (Actual); Status verified 2024-03

CONDITIONS: Metastatic Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — abemaciclib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- 200 mg Abemaciclib With a Meal (Experimental): 200 mg abemaciclib given twice a day (BID) orally with a meal.
  Interventions: Drug: Abemaciclib
- 200 mg Abemaciclib Without a Meal (Experimental): 200 mg abemaciclib given twice a day (BID) orally without a meal, taken in the modified fasted condition.
  Interventions: Drug: Abemaciclib
- 200 mg Abemaciclib Without Regard to Food (Experimental): 200 mg abemaciclib given twice a day (BID) orally without regard for food.
  Interventions: Drug: Abemaciclib

INTERVENTIONS:
Drug: Abemaciclib — Administered orally.
  Other Names: LY2835219

SUMMARY:
The main purpose of this study is to examine the side effects that participants with metastatic breast cancer experience when taking abemaciclib with or without food.

ELIGIBILITY:
Inclusion Criteria:

* Have a diagnosis of HR+, HER2- metastatic breast cancer (mBC).
* Have all of the following:

  * Recurrent, locally advanced, unresectable or mBC with disease progression following anti-estrogen therapy.
  * Prior treatment with chemotherapy for locally advanced or metastatic disease.
  * No prior treatment with cyclin-dependent kinases (CDK) 4 and 6 inhibitor.
* Have Eastern Cooperative Oncology Group performance status (ECOG PS) ≤1.
* Have discontinued all previous treatments for cancer and recovered from the acute effects of therapy.
* Have adequate organ function.
* Women of child-bearing potential must have a negative pregnancy test.
* Are able to swallow tablets/capsules.

Exclusion Criteria:

* Are currently receiving treatment in a clinical study involving an investigational product.
* Have a serious concomitant systemic disorder.
* Have symptomatic central nervous system (CNS) malignancy or metastasis.
* Have a symptomatic Human Immunodeficiency Virus (HIV) infection or symptomatic activated/reactivated hepatitis A, B, or C.
* Have a personal history of syncope of either unexplained or cardiovascular etiology, ventricular tachycardia, ventricular fibrillation, or sudden cardiac arrest.
* Have a history of any other cancer.
* Had major surgery within 14 days prior to randomization.
* Are breastfeeding.
* Have received treatment with a drug that has not received regulatory approval for any indication within 14 or 21 days of the initial dose of study drug for a nonmyelosuppressive or myelosuppressive agent, respectively.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2018-11-28 (Actual); Primary Completion 2019-07-29 (Actual); Study Completion 2023-03-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (15):
- Australia (4):
  - Mater Private Hospital, North Sydney, New South Wales
  - St Vincent's Hospital, Sydney, New South Wales
  - Ashford Cancer Centre Research, Kurralta Park, South Australia
  - Peter MacCallum Cancer Centre, Melbourne, Victoria
- Universitaire Ziekenhuizen Leuven - Campus Gasthuisberg, Leuven, Belgium
- Russia (2):
  - Russian Oncological Research Center, Moscow
  - Volgograd regional clinical oncology dispensary, Volgograd
- Spain (4):
  - Hospital Quirón Salud Barcelona-Instituto Oncológico Baselga, Barcelona
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital Ruber Internacional, Madrid
  - Hospital Clinico San Carlos, Madrid
- Turkey (Türkiye) (4):
  - Akdeniz University Medical Faculty, Antalya
  - Trakya University Faculty of Medicine, Edirne
  - Medical Park Izmir Hospital, Izmir
  - Inonu University Medical Faculty, Malatya

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and EU, whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: https://vivli.org/

REFERENCES:
- See also: A Study of Abemaciclib (LY2835219) With and Without Food in Participants With Metastatic Breast Cancer — https://trials.lilly.com/en-US/trial/184954

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | 200 mg Abemaciclib With a Meal | 200 mg Abemaciclib Without a Meal | 200 mg Abemaciclib Without Regard to Food
Started | 24 | 24 | 24
Received at Least One Dose of Study Drug | 24 | 23 | 24
Completed (Study completers are participants who completed 3 cycles of study treatment (28-day cycle)) | 20 | 18 | 22
Not Completed | 4 | 6 | 2
Not completed — Death | 2 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 3 | 0
Not completed — Completed < 3 Cycles | 2 | 2 | 2

BASELINE CHARACTERISTICS:
Population: All randomized participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | 200 mg Abemaciclib With a Meal | 200 mg Abemaciclib Without a Meal | 200 mg Abemaciclib Without Regard to Food | Total
Number analyzed (Participants) | 24 | 24 | 24 | 72
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.2 (11.6) | 56.9 (11.1) | 57.6 (8.3) | 57.6 (10.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 24 | 24 | 71
  Male | 1 | 0 | 0 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 1 | 1
  Not Hispanic or Latino | 24 | 19 | 20 | 63
  Unknown or Not Reported | 0 | 5 | 3 | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 2 | 0 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 22 | 24 | 24 | 70
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Turkey | 6 | 6 | 6 | 18
  Belgium | 0 | 1 | 0 | 1
  Australia | 11 | 10 | 10 | 31
  Spain | 6 | 6 | 7 | 19
  Russia | 1 | 1 | 1 | 3

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Severe Diarrhea (≥ Grade 3)
Description: Percentage of participants with severe diarrhea (≥ grade 3) during the first 3 cycles. Events were as assessed by the investigator and graded according to Common Terminology Criteria for Adverse Events (CTCAE). Grade 3 was defined as an increase of ≥7 stools per day over baseline; incontinence; hospitalization indicated; severe increase in ostomy output compared to baseline; limiting self-care activities of daily living (ADL).
Time Frame: Cycle 3 (28 Days Cycle)
Population: All participants who received at least one dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | 200 mg Abemaciclib With a Meal | 200 mg Abemaciclib Without a Meal | 200 mg Abemaciclib Without Regard to Food
Number analyzed (Participants) | 24 | 23 | 24
percentage of participants | 4.2 | 0 | 0

2. Primary Outcome: Percentage of Participants With Prolonged Grade 2 Diarrhea
Description: Percentage of participants with prolonged grade 2 diarrhea during first 3 cycles. Events were as assessed by the investigator and graded according to Common Terminology Criteria for Adverse Events (CTCAE). Prolonged Grade 2 diarrhea was any event lasting more than 7 days. Grade 2 was defined as Increase of 4-6 stools per day over baseline; moderate increase in ostomy output compared to baseline.
Time Frame: Cycle 3 (28 Days Cycle)
Population: All participants who received at least one dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | 200 mg Abemaciclib With a Meal | 200 mg Abemaciclib Without a Meal | 200 mg Abemaciclib Without Regard to Food
Number analyzed (Participants) | 24 | 23 | 24
percentage of participants | 8.3 | 17.4 | 20.8

3. Primary Outcome: Percentage of Participants With Dose Reductions Due to Diarrhea
Description: Percentage of participants with dose reductions due to diarrhea during first 3 cycles.
Time Frame: Cycle 3 (28 Days Cycle)
Population: All participants who received at least one dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | 200 mg Abemaciclib With a Meal | 200 mg Abemaciclib Without a Meal | 200 mg Abemaciclib Without Regard to Food
Number analyzed (Participants) | 24 | 23 | 24
percentage of participants | 16.7 | 8.7 | 12.5

4. Primary Outcome: Percentage of Participants With Dose Interruptions Due to Diarrhea
Description: Percentage of participants with dose interruptions due to diarrhea during first 3 cycles.
Time Frame: Cycle 3 (28 Days Cycle)
Population: All participants who received at least one dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | 200 mg Abemaciclib With a Meal | 200 mg Abemaciclib Without a Meal | 200 mg Abemaciclib Without Regard to Food
Number analyzed (Participants) | 24 | 23 | 24
percentage of participants | 16.7 | 4.3 | 8.3

5. Primary Outcome: Percentage of Participants Who Discontinue Treatment Due to Diarrhea
Description: Percentage of participants who discontinue treatment due to diarrhea
Time Frame: Cycle 3 (28 Days Cycle)
Population: All participants who received at least one dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | 200 mg Abemaciclib With a Meal | 200 mg Abemaciclib Without a Meal | 200 mg Abemaciclib Without Regard to Food
Number analyzed (Participants) | 24 | 23 | 24
percentage of participants | 0 | 0 | 0

6. Primary Outcome: Percentage of Participants Utilizing Antidiarrheals
Description: Percentage of participants who utilized anti diarrheals at least once during the first 3 cycles.
Time Frame: Cycle 3 (28 Days Cycle)
Population: All participants who received at least one dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | 200 mg Abemaciclib With a Meal | 200 mg Abemaciclib Without a Meal | 200 mg Abemaciclib Without Regard to Food
Number analyzed (Participants) | 24 | 23 | 24
percentage of participants | 95.8 | 91.3 | 95.8

7. Secondary Outcome: Pharmacokinetics (PK): Mean Steady State Exposure of Abemaciclib
Description: PK: Mean steady state exposure of abemaciclib
Time Frame: Cycle 1: Day 15; Cycle 2: Day 1, Day 15; Cycle 3: Day 1 (28 Days Cycle)
Population: All participants who received at least one dose of study drug who had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram/milliliter (ng/mL)
Arm/Group | 200 mg Abemaciclib With a Meal | 200 mg Abemaciclib Without a Meal | 200 mg Abemaciclib Without Regard to Food
Number analyzed (Participants) | 24 | 21 | 21
nanogram/milliliter (ng/mL)
  Cycle 1: Day 15: number analyzed (Participants) | 23 | 16 | 21
  Cycle 1: Day 15 | 305 (198) | 369 (64) | 356 (75)
  Cycle 2: Day 1: number analyzed (Participants) | 15 | 12 | 18
  Cycle 2: Day 1 | 320 (91) | 280 (99) | 190 (284)
  Cycle 2: Day 15: number analyzed (Participants) | 14 | 13 | 15
  Cycle 2: Day 15 | 77.4 (731) | 345 (51) | 223 (250)
  Cycle 3: Day 1: number analyzed (Participants) | 10 | 13 | 14
  Cycle 3: Day 1 | 135 (896) | 330 (54) | 85.4 (498)

8. Secondary Outcome: PK: Mean Steady State Exposure of Abemaciclib Metabolite LSN2839567
Description: PK: Mean steady state exposure of abemaciclib metabolite LSN2839567
Time Frame: Cycle 1: Day 15; Cycle 2: Day1, Day 15; Cycle 3: Day 1 (28 Days Cycle)
Population: All participants who received at least one dose of study drug who had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram/milliliter (ng/mL)
Arm/Group | 200 mg Abemaciclib With a Meal | 200 mg Abemaciclib Without a Meal | 200 mg Abemaciclib Without Regard to Food
Number analyzed (Participants) | 24 | 21 | 21
nanogram/milliliter (ng/mL)
  Cycle 1 Day 15: number analyzed (Participants) | 23 | 16 | 21
  Cycle 1 Day 15 | 139 (109) | 129 (48) | 159 (61)
  Cycle 2 Day 1: number analyzed (Participants) | 15 | 12 | 19
  Cycle 2 Day 1 | 125 (62) | 109 (84) | 96.3 (127)
  Cycle 2 Day 15: number analyzed (Participants) | 14 | 13 | 15
  Cycle 2 Day 15 | 50.4 (276) | 121 (45) | 112 (79)
  Cycle 3 Day 1: number analyzed (Participants) | 10 | 13 | 14
  Cycle 3 Day 1 | 89.4 (110) | 125 (48) | 61.7 (122)

9. Secondary Outcome: PK: Mean Steady State Exposure of Abemaciclib Metabolite LSN3106726
Description: PK: Mean steady state exposure of abemaciclib metabolite LSN3106726
Time Frame: Cycle 1: Day 15; Cycle 2: Day1, Day 15; Cycle 3: Day 1 (28 Days Cycle)
Population: All participants who received at least one dose of study drug who had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram/milliliter (ng/mL)
Arm/Group | 200 mg Abemaciclib With a Meal | 200 mg Abemaciclib Without a Meal | 200 mg Abemaciclib Without Regard to Food
Number analyzed (Participants) | 24 | 21 | 21
nanogram/milliliter (ng/mL)
  Cycle 1 Day 15: number analyzed (Participants) | 23 | 16 | 21
  Cycle 1 Day 15 | 231 (120) | 242 (38) | 287 (63)
  Cycle 2 Day 1: number analyzed (Participants) | 15 | 12 | 19
  Cycle 2 Day 1 | 230 (59) | 210 (57) | 152 (222)
  Cycle 2 Day 15: number analyzed (Participants) | 14 | 13 | 15
  Cycle 2 Day 15 | 80.5 (377) | 221 (31) | 182 (112)
  Cycle 3 Day 1: number analyzed (Participants) | 10 | 13 | 14
  Cycle 3 Day 1 | 146 (174) | 223 (33) | 107 (172)

ADVERSE EVENTS:
Time Frame: Baseline until end of the follow-up (Up To 44 months)
Description: All participants who received at least one dose of study drug.
Arm/Group | 200 mg Abemaciclib With a Meal | 200 mg Abemaciclib Without a Meal | 200 mg Abemaciclib Without Regard to Food
All-Cause Mortality (participants affected / at risk) | 3/24 | 4/23 | 1/24
Serious Adverse Events (participants affected / at risk) | 3/24 | 5/23 | 8/24
Other Adverse Events (participants affected / at risk) | 24/24 | 23/23 | 24/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 200 mg Abemaciclib With a Meal (N=24) | 200 mg Abemaciclib Without a Meal (N=23) | 200 mg Abemaciclib Without Regard to Food (N=24)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 3 (3) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 2 (2) | 0 (0)
Non-cardiac chest pain (General disorders) | 1 (1) | 0 (0) | 0 (0)
Cholangitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Hepatic function abnormal (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Cauda equina syndrome (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Guillain-barre syndrome (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Renal failure (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Superficial vein thrombosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 200 mg Abemaciclib With a Meal (N=24) | 200 mg Abemaciclib Without a Meal (N=23) | 200 mg Abemaciclib Without Regard to Food (N=24)
Anaemia (Blood and lymphatic system disorders) | 14 (34) | 11 (19) | 10 (33)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (5) | 1 (2)
Lymphopenia (Blood and lymphatic system disorders) | 2 (3) | 1 (3) | 2 (3)
Neutropenia (Blood and lymphatic system disorders) | 6 (18) | 8 (21) | 9 (25)
Pancytopenia (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 2 (4) | 2 (2)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Ear pain (Ear and labyrinth disorders) | 1 (1) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1)
Cushingoid (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1)
Hyperthyroidism (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0)
Dry eye (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Lacrimation increased (Eye disorders) | 2 (3) | 2 (2) | 2 (8)
Lid sulcus deepened (Eye disorders) | 0 (0) | 0 (0) | 1 (5)
Vision blurred (Eye disorders) | 0 (0) | 0 (0) | 2 (9)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 2 (2) | 2 (2) | 1 (4)
Abdominal pain (Gastrointestinal disorders) | 10 (12) | 4 (5) | 5 (8)
Abdominal pain upper (Gastrointestinal disorders) | 2 (3) | 2 (3) | 2 (4)
Angular cheilitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Ascites (Gastrointestinal disorders) | 0 (0) | 1 (2) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1) | 1 (1) | 3 (3)
Diarrhoea (Gastrointestinal disorders) | 21 (204) | 22 (187) | 22 (229)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 4 (12)
Flatulence (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 3 (3) | 1 (1) | 1 (1)
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Mallory-weiss syndrome (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Mouth ulceration (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 15 (16) | 11 (21) | 14 (20)
Odynophagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Oral blood blister (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Retching (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2)
Toothache (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 10 (23) | 10 (20) | 7 (10)
Asthenia (General disorders) | 6 (10) | 5 (12) | 4 (12)
Chest pain (General disorders) | 1 (1) | 1 (1) | 0 (0)
Fatigue (General disorders) | 11 (15) | 4 (5) | 10 (20)
Ill-defined disorder (General disorders) | 0 (0) | 0 (0) | 1 (1)
Malaise (General disorders) | 1 (1) | 0 (0) | 0 (0)
Mucosal dryness (General disorders) | 0 (0) | 0 (0) | 1 (1)
Mucosal inflammation (General disorders) | 3 (3) | 1 (1) | 5 (6)
Nodule (General disorders) | 0 (0) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 1 (3) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 2 (2) | 2 (2)
Pyrexia (General disorders) | 2 (2) | 2 (2) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Hepatic failure (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Hepatic pain (Hepatobiliary disorders) | 1 (1) | 0 (0) | 1 (1)
Hepatomegaly (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Hypertransaminasaemia (Hepatobiliary disorders) | 1 (1) | 0 (0) | 1 (1)
Seasonal allergy (Immune system disorders) | 0 (0) | 1 (1) | 0 (0)
Bacterial rhinitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Conjunctivitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Covid-19 (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Dermatophytosis of nail (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Diverticulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Oral herpes (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Paronychia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 1 (2) | 1 (1) | 0 (0)
Pyelonephritis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
Rhinitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0) | 1 (2)
Skin bacterial infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Tinea pedis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Tooth infection (Infections and infestations) | 0 (0) | 1 (2) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 4 (6) | 0 (0) | 3 (3)
Urinary tract infection (Infections and infestations) | 4 (4) | 2 (2) | 2 (2)
Viral infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Viral upper respiratory tract infection (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Vulvovaginal candidiasis (Infections and infestations) | 1 (2) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 3 (4) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (2) | 0 (0) | 0 (0)
Spinal fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 4 (7) | 2 (3) | 5 (9)
Aspartate aminotransferase increased (Investigations) | 6 (11) | 4 (7) | 4 (8)
Blood alkaline phosphatase increased (Investigations) | 2 (4) | 2 (2) | 4 (8)
Blood bilirubin increased (Investigations) | 3 (3) | 3 (7) | 1 (1)
Blood calcium decreased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Blood creatinine decreased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Blood creatinine increased (Investigations) | 3 (4) | 5 (10) | 4 (8)
Blood lactate dehydrogenase decreased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Blood lactate dehydrogenase increased (Investigations) | 0 (0) | 2 (3) | 0 (0)
Blood phosphorus decreased (Investigations) | 1 (1) | 1 (2) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 3 (5) | 4 (7) | 4 (10)
Glomerular filtration rate decreased (Investigations) | 0 (0) | 0 (0) | 1 (2)
Haemoglobin decreased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Hepatic enzyme increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Lymphocyte count decreased (Investigations) | 5 (19) | 3 (6) | 5 (20)
Neutrophil count decreased (Investigations) | 7 (35) | 6 (15) | 10 (41)
Platelet count decreased (Investigations) | 11 (34) | 7 (16) | 5 (12)
Protein total decreased (Investigations) | 0 (0) | 1 (3) | 0 (0)
Weight decreased (Investigations) | 2 (2) | 5 (7) | 3 (4)
White blood cell count decreased (Investigations) | 9 (31) | 7 (27) | 7 (39)
Decreased appetite (Metabolism and nutrition disorders) | 8 (11) | 8 (12) | 9 (11)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hyperuricaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 2 (4) | 3 (10) | 1 (2)
Hypocalcaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (2) | 1 (2)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (2) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 5 (8) | 2 (4)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 2 (3) | 0 (0)
Hypophosphataemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 2 (2)
Vitamin b12 deficiency (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (4) | 4 (4)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (4) | 0 (0) | 5 (6)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Groin pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Joint stiffness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Limb discomfort (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Sacral pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2)
Tendonitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Metastases to meninges (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Balance disorder (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Brain fog (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Disturbance in attention (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 5 (6) | 2 (2) | 1 (1)
Dysgeusia (Nervous system disorders) | 2 (2) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 5 (7) | 2 (2) | 0 (0)
Hemiparesis (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Lethargy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Memory impairment (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Sensory disturbance (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Sensory loss (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Sleep deficit (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 1 (1) | 2 (2)
Taste disorder (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Affect lability (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Depressed mood (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (1)
Insomnia (Psychiatric disorders) | 2 (2) | 0 (0) | 0 (0)
Dysuria (Renal and urinary disorders) | 1 (1) | 1 (1) | 0 (0)
Hydronephrosis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Nocturia (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 5 (6) | 1 (1)
Dry throat (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 1 (1) | 1 (1)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (2) | 3 (3)
Dry skin (Skin and subcutaneous tissue disorders) | 2 (3) | 1 (1) | 1 (1)
Nail ridging (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Onychoclasis (Skin and subcutaneous tissue disorders) | 2 (3) | 0 (0) | 0 (0)
Onychomadesis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Pain of skin (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 4 (6) | 3 (3)
Rash (Skin and subcutaneous tissue disorders) | 4 (4) | 2 (3) | 2 (2)
Rash macular (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Abdominal cavity drainage (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
Tooth extraction (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Hot flush (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 1 (1) | 1 (2)
Lymphoedema (Vascular disorders) | 0 (0) | 0 (0) | 1 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2020-02-10): https://cdn.clinicaltrials.gov/large-docs/66/NCT03703466/Prot_000.pdf
  • Statistical Analysis Plan (2018-11-08): https://cdn.clinicaltrials.gov/large-docs/66/NCT03703466/SAP_001.pdf